CLINICAL TRIAL: NCT00105703
Title: Evaluation of a Nurse Case Management Model for Chronic Heart Failure
Acronym: CHF ENCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHI 99-236
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-09

CONDITIONS: Heart Failure, Congestive
Keywords: Nurse practitioners; Case management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Case management using advanced nurse practitioners

INTERVENTIONS:
Behavioral: Case management using advanced nurse practitioners

SUMMARY:
Despite established clinical practice guidelines, wide variations exist in the care of chronic heart failure (CHF) patients in Veterans Health Administration. Previous randomized, controlled studies have suggested that a nurse case management model may improve the outcomes of care for patients with CHF. However, these studies involved selected groups of patients (i.e., those who agreed to participate in randomized trials) in selected settings (i.e., tertiary care facilities); so, the findings are not likely to be indicative of the true effectiveness of case management in a large population of CHF patients.

DETAILED DESCRIPTION:
BACKGROUND / RATIONALE:

Despite established clinical practice guidelines, wide variations exist in the care of chronic heart failure (CHF) patients in Veterans Health Administration. Previous randomized, controlled studies have suggested that a nurse case management model may improve the outcomes of care for patients with CHF. However, these studies involved selected groups of patients (i.e., those who agreed to participate in randomized trials) in selected settings (i.e., tertiary care facilities); so, the findings are not likely to be indicative of the true effectiveness of case management in a large population of CHF patients.

OBJECTIVE(S):

This study will evaluate the impact of a nurse practitioner case management model compared with usual care in patients with congestive heart failure (CHF). Outcomes include health-related quality of life, patient satisfaction, compliance with medication guidelines, mortality, readmissions, bed days of care, outpatient visits, emergency room visits, and pharmacy costs.

METHODS:

Patients with CHF will be identified by review of admission/discharge logs, review of clinic schedules, and referrals from medical personnel. All patients in the northern half of VISN 11 (Ann Arbor, Detroit, Saginaw, and Battle Creek) will participate in a case management program, in which they will receive care from nurse practitioners who will be supported by practice guidelines, treatment algorithms, and guidance from cardiologists at the VA Ann Arbor Health Care System. Patients in the southern half of the VISN (Indianapolis and Danville) will make up the comparison group and will receive usual care for CHF patients.

All study participants will complete baseline and one and two year follow-up questionnaires on health related quality of life, including the SF-36V and the Minnesota Living With Heart Failure Questionnaire. Patient satisfaction will be assessed using the VA National Ambulatory Care Survey. Additional data on the use of health care resources over the two years following each patient�s index hospitalization will be collected from the Patient Treatment File (PTF) and the Outpatient Census (OPC) File. Data on compliance with medication guidelines will be obtained from the VISN 11 pharmacy database. Multivariate analyses will be used, with the main study outcomes as dependent variables and intervention vs. comparison group membership as independent variables, controlling for baseline differences between intervention and comparison groups. Additional analyses will compare the study outcomes for patients served by primary versus tertiary sites.

Semi-structured interviews will be conducted with participating providers at the beginning, middle, and end of the study, to determine satisfaction with the program, as well as specific components that were perceived to help or hinder its effectiveness.

STATUS:

All two-year follow-up questionnaires have been received and entered. Medical record abstraction, which includes data on severity of disease, will continue through Dec 2007. All interviews with medical center staff have been conducted, transcribed, and coded. We are in the process of pulling one-year prior and one and two-year post data on comorbidities and resource utilization. Analysis of survey, medical record, interview, and secondary data will continue through spring of 2008, when the final report will be written.

ELIGIBILITY:
Inclusion Criteria:

* Patient receives all cardiology care at a VISN 11 VAMC.
* Must have chronic heart failure (CHF) secondary to systolic or diastolic dysfunction, as defined by meeting (1) or (2) below:

  1. Systolic Dysfunction, defined by a history or documentation of LVEF = 40% (or fractional shortening = 20%-if LVEF not documented)

     AND at least ONE of the following:
     * Current diagnosis or history of CHF and/or
     * Physical findings and/or symptoms of CHF within two months of enrollment and/or
     * Hospitalization for CHF within 12 months OR
  2. Diastolic Dysfunction, defined by a history of documentation of LVEF > 40% (or fractional shortening > 20% if LVEF not documented) AND Physical findings and/or symptoms of CHF within two months of enrollment.

Exclusion Criteria:

Based on medical record data, patient does not have any co-morbidity other than CHF which, in the opinion of the investigator, limits life expectancy to less than six months (e.g., metastatic CA, hospice care, renal failure with a creatinine above 5.0 mg/dL or on dialysis, HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 969 (Actual)
Dates: Start 2002-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The following outcomes will be measured at one and two years following each participant's enrollment in the study: mortality, health related quality of life, patient satisfaction with care, resource utilization (outpatient visits, admissions.

SECONDARY OUTCOMES:
Feedback regarding the intervention from the directors, chiefs of staff, cardiologists, nurse practitioners, and primary care providers at the participating sites.

CONTACTS AND LOCATIONS:
Overall Officials: Julie C Lowery, PhD MHSA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (4):
- United States (4):
  - VA Illiana Health Care System, Danville, IL, Danville, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan

REFERENCES:
- [Result] Subramanian U, Weinberger M, Eckert GJ, L'Italien GJ, Lapuerta P, Tierney W. Geographic variation in health care utilization and outcomes in veterans with acute myocardial infarction. J Gen Intern Med. 2002 Aug;17(8):604-11. doi: 10.1046/j.1525-1497.2002.11048.x. PMID 12213141
- [Result] Subramanian U, Sutherland J, Hopp F, Lowery J, Doebbeling B. Patient self-efficacy, provider self-management counseling and health status among patients with chronic heart failure. Journal of general internal medicine. 2005 Oct 1; 20(Supplement 1):70.
- [Result] Subramanian U, Weinberger M, Fihn SD, Tierney WM. Diagnostic challenges defining heart failure when using echocardiograms. Am J Cardiol. 2003 Apr 15;91(8):1015-7, A8. doi: 10.1016/s0002-9149(03)00130-9. No abstract available. PMID 12686354
- [Result] Subramanian U, Hopp F, Mitchinson A, Lowery J. Impact of provider self-management education, patient self-efficacy, and health status on patient adherence in heart failure in a Veterans Administration population. Congest Heart Fail. 2008 Jan-Feb;14(1):6-11. doi: 10.1111/j.1751-7133.2008.07174.x. PMID 18256563
- See also: Ann Arbor HSR&D Center of Excellence Web page — http://www.annarbor.hsrd.research.va.gov/